CLINICAL TRIAL: NCT05095753
Title: Data Collection of Heart Rate and Blood Pressure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: MindMics Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: 120190480
Record Dates: First submitted 2021-10-07; First posted 2021-10-27 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Healthy People

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Earbud — In ear headphone with embedded infrasonic hemodynography technology

SUMMARY:
The purpose of the study is data collection for building and validating the algorithms for analytics of vital signs using wearable earphones (MindMics device).

DETAILED DESCRIPTION:
MindMics is developing technology to enhance an individual's quality of life by continuously monitoring the heart rate, stress thereby allowing people to make better decisions regarding their health. MindMics has a working prototype of the ear buds which will perform all the conventional tasks earbuds do (listen to music, etc.), but, in addition, will measure your vital signs. The earbuds capture the sounds made by the various cardiac structures pulsing and moving blood.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-90
* No gender restrictions
* Cognitive ability to consent

Exclusion Criteria:

* Patients with pacemakers
* Patients with irregular heart rhythms

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Healthy cohort
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-11-15 (Actual); Primary Completion 2021-11-14 (Estimated); Study Completion 2021-11-14 (Estimated)

PRIMARY OUTCOMES:
RR Interval from ECG signal | 20 minutes
  Time in milliseconds between successive ECG R peaks
Inter-beat Interval from earbud signal | 20 minutes
  Time in milliseconds between successive peaks in earbud signal
Systolic and diastolic blood pressure from blood pressure cuff | 20 minutes
  Value of blood pressure in mmHg reported by a blood pressure cuff

CONTACTS AND LOCATIONS:
Locations (1):
- MindMics, Inc., Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
No plan.